CLINICAL TRIAL: NCT05726461
Title: Efficacy and Safety of Android Artificial Pancreas System Use at Home Among Type 1 Diabetes Mellitus Adults in China: Protocol of a 26-Week, Free-Living, Randomized, Open-Label, Two-Arm, Two-Phase, Crossover Trial
Brief Title: Efficacy and Safety of Android Artificial Pancreas System in Adult Patients With Type 1 Diabetes Mellitus in China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jinhua Yan, Vice Professor,Principal Investigator,Department of Endocrinology and Metabolism, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MLei
Record Dates: First submitted 2023-01-18; First posted 2023-02-14 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Metabolic Disease; Endocrine System Diseases; Autoimmune Diseases; Immune System Diseases
Keywords: Type 1 diabetes mellitus;; Artificial pancreas system;; Do-it-yourself artificial pancreas system;; Automated insulin delivery;; Hybrid closed loop;; Adult; AndroidAPS
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Autoimmune Diseases; Immune System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AndroidAPS-rt-CGM (Experimental): 1) AiDEX G7 continuous glucose monitoring (an rt-CGM);2) Equil® insulin patch pump;3) AndroidAPS algorithm implemented in Android smartphone
  Interventions: Device: AndroidAPS-rt-CGM;
- sensor augmented pump(SAP) (Active Comparator): SAP includes only Equil® insulin patch pump and AiDEX G7 continuous glucose monitoring.
  Interventions: Device: sensor augmented pump(SAP);

INTERVENTIONS:
Device: AndroidAPS-rt-CGM; — Insulin therapy (aspart, lispro or glulisine) with AndroidAPS-rt-CGM.AndroidAPS-rt-CGM consists of three components:1) AiDEX G7 continuous glucose monitoring (an rt-CGM);2) Equil® insulin patch pump;3) AndroidAPS algorithm implemented in Android smartphone.
  Arms: AndroidAPS-rt-CGM
Device: sensor augmented pump(SAP); — Insulin therapy (aspart, lispro or glulisine) with sensor augmented pump(SAP).SAP includes only Equil® insulin patch pump and AiDEX G7 continuous glucose monitoring.
  Arms: sensor augmented pump(SAP)

SUMMARY:
This is a 26-week randomized, free-living, open-label, two-arm, two-phase, crossover trial. Participants will receive two interventions at different phases, including the Android artificial pancreas system(AndroidAPS-rt-CGM) and sensor-augment pump(SAP), and use marketed rapid-acting insulin analogs (insulin Aspart, insulin Lispro, or insulin Glulisine) normally used in their usual clinical care. The safety and efficacy of AndroidAPS-rt-CGM and SAP in adult T1DM with suboptimal glycemic control will be compared to explore whether the use of AndroidAPS-rt-CGM in adult T1DM with suboptimal glycemic control will be associated with better glycemic control with no increased hypoglycemia.

DETAILED DESCRIPTION:
All participants will be free to live during the study. Each intervention phase is 12 weeks, preceded by a 2-week training period and separated by a 2-week washout period. During the training period, eligible participants will be trained to use the study rt-CGM and insulin pump and randomly assigned 1:1 to two treatment sequences after the training period. In Sequence A, patients use AndroidAPS-rt-CGM for the first intervention period (phase 1) and SAP for the second intervention period (phase 2); in Sequence B, patients use SAP for Phase 1 and AndroidAPS-rt-CGM for Phase 2. Participants who enter sequences A and B will be trained to use the study devices running in automated insulin delivery(AID) mode on the first day of phase 1 and phase 2, respectively. AndroidAPS-rt-CGM consists of three components:1) AiDEX G7 continuous glucose monitoring (an rt-CGM);2) Equil® insulin patch pump;3) AndroidAPS algorithm implemented in Android smartphone. The participants will use the study patch pump and rt-CGM, but the AndroidAPS algorithm and advanced features will not be allowed during the SAP intervention period. During the washout period, participants will continue using the study insulin pump with their standard settings, but the study rt-CGM will be replaced by daily self-monitoring of fingerstick glucose. The primary endpoint is time in range (3.9-10.0 mmol/L) derived from CGM. The main secondary endpoints include the percentage of sensor glucose values below, within, and above the target range; mean sensor glucose value; measures of glycemic variability, and centralized HbA1c. Safety endpoints mainly include the frequency of hypoglycemia events, diabetic ketoacidosis, and other serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

Prior to this study:

1. Type 1 diabetes mellitus(T1DM) was diagnosed by an endocrinologist for at least one year.
2. Aged from 18 to 75 years.
3. HbA1c was 7.0% ~ 11%.
4. on multiple daily injection(MDI) or insulin pump therapy for ≥3 months with less than 20% insulin dose changes.
5. The total daily dose(TDD) were≥0.3 u/kg /day, and the basal rate was ≥0.05 u/hour.
6. Regular self-monitoring of blood glucose (≥3 times per day) for ≥2 months.
7. Lived with an adult willing to care for the subject during the study.
8. Women of childbearing age are willing to use appropriate contraceptive measures.
9. Willing to follow the research protocol.
10. Have daily access to a Wi-Fi network.

Exclusion Criteria:

Prior to this study:

1. Severe acute or chronic complications of diabetes mellitus.
2. Frequent severe hypoglycemia in the past three months.
3. Patients who have used closed-loop therapy in the last two months (excluding those who have recently used CGM) and those participating in other studies.
4. Abnormal liver function (ALT was 2.5 times higher than the upper limit of normal).
5. Moderate to severe renal impairment (eGFR<60ml/min/1.73m2).
6. Clinically significant heart disease.
7. Pregnant or planning pregnancy.
8. Used drugs that can interfere with glucose metabolism (e.g., exogenous glucocorticoids, nonselective beta-blockers, monoamine oxidase inhibitors) in the past eight weeks.
9. Frequent acetaminophen, drug abuse, and excessive drinking.
10. Known allergy to medical-grade adhesives or CGM and its affiliated components.
11. Severe visual or hearing impairment.
12. Severe skin disease at the site of sensor implantation.
13. Plan to undergo elective surgery requiring general anesthesia during the study.
14. Eating disorders such as anorexia or bulimia.
15. Other physical or psychological conditions deemed inappropriate for inclusion by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-02-11 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Time in range(TIR) | during the last 2 weeks of each phase
  TIR(3.9-10.0 mmol/l) derived from CGM will be collected during the last 2 weeks of each phase.

SECONDARY OUTCOMES:
Glycosylated Hemoglobin A1c(HbA1c) | on the last day of each phase
  centralized HbA1c will be measured on the last day of each phase
Time in target range(TIT) | during the last 2 weeks of each phase.
  TIT(3.9-7.8 mmol/l) derived from CGM will be collected during the last 2 weeks of each phase.
Time above range(TAR) | during the last 2 weeks of each phase.
  TAR(> 10.0 mmol/L and > 13.9 mmol/L) derived from CGM will be collected during the last 2 weeks of each phase.
Time below range(TBR) | during the last 2 weeks of each phase.
  TBR(< 3.9 mmol/L and <3.0 mmol/L) derived from CGM will be collected during the last 2 weeks of each phase.
Mean blood glucose value(MBG) | during the last 2 weeks of each phase.
  MBG derived from CGM will be collected during the last 2 weeks of each phase.
Standard deviation(SD) | during the last 2 weeks of each phase.
  SD derived from CGM will be collected during the last 2 weeks of each phase.
Coefficient of variation(CV) | during the last 2 weeks of each phase.
  CV derived from CGM will be collected during the last 2 weeks of each phase.
Mean amplitude of glucose excursions(MAGE) | during the last 2 weeks of each phase.
  MAGE derived from CGM will be collected during the last 2 weeks of each phase.
the Chinese version of Hypoglycemia Fear Survey II-Worry Scale(HFS-II) | in week 0 ,week 12, week 14, and week 26
  The Chinese version of Hypoglycemia Fear Survey II- Worry Scale is used to evaluate the psychological status of diabetic patients. Change in Hypoglycemia Fear Scale (HFS) score will be assessed in week 12 and week 26 adjusted for baseline(week 0 and week 14). These validated surveys include 18 questions to measure hypoglycemia-related anxiety and fear. Each item is rated on a 5-point Likert scale from 0(never related) to 4(very related). "Never relative" scores 1, " and "very related" scores 4. Patients with higher scores are considered with more anxiety and fear of hypoglycemia. The change in HFS-II will be assessed in week 12 and week 26 adjusted for baseline(weeks 0 and 14).
Frequency of hypoglycemia events | 12 weeks for each arm of the crossover
  Level 1 is defined as sensor glucose ≤3.9mmol/L;level 2 is defined as sensor glucose ≤3.0mmol/L; level 3 is defined as hypoglycemia accompanied by severe cognitive impairment requiring the assistance of another individual to administer rescue therapy.
Frequency of diabetic ketoacidosis (DKA) | 12 weeks for each arm of the crossover
  DKA can be diagnosed when the following three points are met: 1)plasma glucose level ≥13.9mmol/L;2)pH<7.3 or bicarbonate <18 mmol/L;3)serum ketone ≥3mmol/L or urine ketone≥2+.
Frequency of serious adverse events about device | 12 weeks for each arm of the crossover
  Serious adverse device effect(ADE) is defined as an event related to the use of the study device which is fatal or life-threatening, resulting in persistent or substantial disability, or requires (or prolonged) hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Jinhua Yan, phD, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University; Wen Xu, phD,MD, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Jinhua Yan, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang Q, Ni Y, Lei M, Ling P, Yan J, Guo X, Yang D, Wang C. Experiences and opinions of adults with type 1 diabetes on the android-based open-source closed-loop system in China: a qualitative study. BMJ Open. 2025 Jan 15;15(1):e094333. doi: 10.1136/bmjopen-2024-094333. PMID 39819904
- [Derived] Lei M, Lin B, Ling P, Liu Z, Yang D, Deng H, Yang X, Lv J, Xu W, Yan J. Efficacy and safety of Android artificial pancreas system use at home among adults with type 1 diabetes mellitus in China: protocol of a 26-week, free-living, randomised, open-label, two-arm, two-phase, crossover trial. BMJ Open. 2023 Aug 9;13(8):e073263. doi: 10.1136/bmjopen-2023-073263. PMID 37558445